CLINICAL TRIAL: NCT01411215
Title: A Non-Interventional Study of the Treatment With Etanercept in Rheumatoid Arthritis (RA) and Ankylosing Spondylitis (AS) Subjects in Rheumatology Department
Brief Title: A Study of Rheumatoid Arthritis Treatment With Enbrel in Adult Patient in Outpatient Department
Acronym: ENBREL NIS CN
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801044
Record Dates: First submitted 2011-05-13; First posted 2011-08-08 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis
Keywords: Rheumatoid arthritis; ankylosing spondylitis; observational study
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA, AS: Rheumatoid arthritis patients Ankylosing spondylitis patients
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: Enbrel — 25mg biweekly or 50mg per week, subcutaneous injection
  Other Names: etanercept

SUMMARY:
This is an open-label, multicenter and observational study in China, which is designed to record the data of RA & AS patients within 52 weeks after rheumatologists decided to prescribe etanercept, and evaluate the safety and efficacy of the treatment. All eligible subjects agreed to be recruited in the study and can withdraw anytime if they choose so.

Patients with RA or AS are typically managed by rheumatologists. As this study seeks to record the data of RA & AS patient in etanercept and evaluate the safety and efficacy of the treatment, patients will be recruited from Rheumatic department. Rheumatologist will be asked to build up the database for RA & AS patient surveillance prospectively in outpatient dept, which benefits for the patient treatment outcomes evaluation and clinical management.

DETAILED DESCRIPTION:
The primary objective of this non-interventional study is to evaluate the safety of etanercept in Chinese RA and AS subjects. Total of 600 subjects (300 RA subjects and 300 AS subjects) will be enrolled in the study. If the true rate of an adverse event is no less than 0.5%, with sample size of 600 subjects, this study will have 95% probability to detect at least one occurrence of the adverse event. The study prematurely discontinued on January 15, 2013 due to slow enrollment and low adherence of etanercept. It should be noted that safety concerns have not been seen in this study and have not factored into this decision.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed diagnosis of rheumatoid arthritis or ankylosing spondylitis.
* Subject has accepted physician's prescription of etanercept in rheumatology department.
* Subject agreed to be enrolled in the observational study and sign the ICD.
* Subject is≥18 years of age at the time of consent.
* Subject is willing and able to understand and complete questionnaires

Exclusion Criteria:

* Presence of active or suspected latent infection including HIV, or any underlying disease, including open cutaneous ulcers that could predispose the subject to infections.
* Immunodeficiency syndromes including Felty syndrome or large granular lymphocyte syndrome.
* Active tuberculosis (TB) or a history of TB, or findings consistent with previous exposure to TB on a chest x-ray (CXR). Investigators must follow China's guidelines for appropriate screening and treatment of TB.
* History of hypersensitivity to any of the ingredients in either preparation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient RA and AS patients in China
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- China (15):
  - Daping Hospital, Chongqing, Chongqing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - No. 199, Haerbin, Heilongjiang
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Jiangsu Province Hospital/Department of Rheumatology, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Si Chuan Huaxi Hospital/Rheumatology Department, Chengdu, Sichuan
  - Baotou Central Hospital, Baotou
  - Shanghai Changning Guanghua Integrative Medicine Hospital, Beijing
  - Shanghai Jiaotong University Affiliated Third People's Hospital, Shanghai
  - Xinjiang Uygur Autonomous Region People's Hospital, Ürümqi

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801044&StudyName=A%20Study%20of%20Rheumatoid%20Arthritis%20Treatment%20with%20Enbrel%20in%20Adult%20Patient%20in%20Outpatient%20Department%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Rheumatoid Arthritis [RA]: Participants with RA who received etanercept 25 mg twice weekly or 50 mg weekly per standard medical practice were observed for 52 weeks
- Ankylosing Spondylitis [AS]: Participants with AS who received etanercept 25 mg twice weekly or 50 mg weekly per standard medical practice were observed for 52 weeks
Period: Overall Study
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Started | 69 | 91
Treated | 69 | 90 (1 participant was considered as screen failure and therefore not treated.)
Completed | 3 | 7
Not Completed | 66 | 84
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 2 | 4
Not completed — Lost to Follow-up | 12 | 18
Not completed — Did not meet entrance criteria | 0 | 1
Not completed — Study terminated by sponsor | 2 | 15
Not completed — Protocol Violation | 3 | 5
Not completed — Withdrawal by Subject | 34 | 21
Not completed — Other | 12 | 17
Not completed — Screen failure | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline participants were all enrolled participants who received at least 1 dose of etanercept.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS] | Total
Number analyzed (Participants) | 69 | 90 | 159
Age, Customized [Number; unit: Participants]
  less than (<) 20 years | 3 | 15 | 18
  greater than or equal to (>=) 20 and <30 years | 3 | 27 | 30
  >=30 and <40 years | 7 | 21 | 28
  >=40 and <50 years | 22 | 18 | 40
  >=50 years | 34 | 9 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 24 | 74
  Male | 19 | 66 | 85

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Any Adverse Events (AEs) During 24 Weeks
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: First day of receiving etanercept through 24 weeks
Population: All enrolled participants who received at least 1 dose of etanercept.
Measure: Number; unit: Participants
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Number analyzed (Participants) | 69 | 90
Participants | 7 | 9

2. Primary Outcome: Number of Participants Who Had Any AEs During 52 Weeks
Description: as for outcome 1
Time Frame: First day of receiving etanercept through 52 weeks
Population: All enrolled participants who received at least 1 dose of etanercept.
Measure: Number; unit: Participants
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Number analyzed (Participants) | 69 | 90
Participants | 8 | 9

3. Primary Outcome: Number of Participants Who Had Any Serious Adverse Events (SAEs) During 24 Weeks
Description: An SAE was defined as an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Informed consent or signed data privacy statement through 24 weeks
Population: All enrolled participants who received at least 1 dose of etanercept.
Measure: Number; unit: Participants
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Number analyzed (Participants) | 69 | 90
Participants | 0 | 0

4. Primary Outcome: Number of Participants Who Had Any SAEs During 52 Weeks
Description: as for outcome 3
Time Frame: Informed consent or signed data privacy statement through 52 weeks
Population: All enrolled participants who received at least 1 dose of etanercept.
Measure: Number; unit: Participants
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Number analyzed (Participants) | 69 | 90
Participants | 0 | 0

5. Primary Outcome: Number of Participants With AEs Per System Organ Class During 24 Weeks
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Participants with multiple AEs within a category (system organ class) were counted once within the category.
Time Frame: First day of receiving etanercept through 24 weeks
Population: All enrolled participants who received at least 1 dose of etanercept.
Measure: Number; unit: Participants
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Number analyzed (Participants) | 69 | 90
Participants
  Eye disorders | 0 | 1
  Gastrointestinal disorders | 0 | 1
  General disorders+administration site conditions | 2 | 1
  Hepatobiliary disorders | 0 | 2
  Infections and infestations | 1 | 1
  Investigations | 3 | 3
  Metabolism and nutrition disorders | 1 | 0
  Musculoskeletal and connective tissue disorders | 0 | 1
  Skin and subcutaneous tissue disorders | 2 | 0

6. Primary Outcome: Number of Participants With AEs Per System Organ Class During 52 Weeks
Description: as for outcome 5
Time Frame: First day of receiving etanercept through 52 weeks
Population: All enrolled participants who received at least 1 dose of etanercept.
Measure: Number; unit: Participants
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Number analyzed (Participants) | 69 | 90
Participants
  Eye disorders | 0 | 1
  Gastrointestinal disorders | 0 | 1
  General disorders+administration site conditions | 2 | 1
  Hepatobiliary disorders | 0 | 2
  Infections and infestations | 1 | 1
  Investigations | 3 | 3
  Metabolism and nutrition disorders | 1 | 0
  Musculoskeletal and connective tissue disorders | 1 | 1
  Skin and subcutaneous tissue disorders | 2 | 0

7. Secondary Outcome: Physician's Global Assessment of Disease Activity
Description: Physicians indicated on a 0-100 millimeters (mm) visual analogue scale (VAS) to assess the activity of the participant's disease according to the participant's clinical condition, with 0 meaning no disease activity (disease inactive) and 100 meaning extreme disease activity (disease extremely active).
Time Frame: Baseline (Week 0), Week 2, Week 4, Week 8, Week 12, Week 24, Week 36, Week 52
Population: All enrolled participants who received at least 1 dose of etanercept. Participants analyzed were participants who were evaluated for physician's global assessment of disease activity. n=number of evaluable participants at the corresponding visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Number analyzed (Participants) | 65 | 82
mm
  Baseline (Week 0), n=65,82 | 63.4 (20.62) | 60.9 (22.91)
  Week 2, n=44,59 | 45.3 (26.33) | 48.2 (29.14)
  Week 4, n=35,61 | 40.5 (30.77) | 44.2 (31.23)
  Week 8, n=24,47 | 34.8 (37.39) | 43.9 (30.76)
  Week 12, n=16,34 | 34.8 (35.22) | 39.2 (35.88)
  Week 24, n=7,18 | 27.4 (35.18) | 30.1 (30.78)
  Week 36, n=2,13 | 5.0 (7.07) | 19.8 (26.49)
  Week 52, n=3,6 | 10.7 (15.14) | 16.5 (12.08)

8. Secondary Outcome: Participant's Global Assessment (PtGA) of Disease Activity
Description: Participants placed a vertical line on a 0-100 mm VAS to indicate the magnitude of their global disease activity, with 0 meaning no disease activity (disease inactive) and 100 meaning extreme disease activity (disease extremely active).
Time Frame: Baseline (Week 0), Week 2, Week 4, Week 8, Week 12, Week 24, Week 36, Week 52
Population: All enrolled participants who received at least 1 dose of etanercept. Participants analyzed were participants who were evaluated for PtGA of disease activity. n=number of evaluable participants at the corresponding visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Number analyzed (Participants) | 65 | 84
mm
  Baseline (Week 0), n=65, 84 | 64.9 (20.27) | 61.8 (21.50)
  Week 2, n=42,61 | 45.1 (27.00) | 48.9 (27.52)
  Week 4, n=35, 60 | 42.2 (31.16) | 44.1 (30.78)
  Week 8, n=23, 47 | 36.1 (38.10) | 44.4 (31.25)
  Week 12, n=16,33 | 34.6 (35.19) | 38.8 (35.54)
  Week 24, n=7,18 | 26.6 (35.02) | 32.1 (32.72)
  Week 36, n=2,12 | 5.0 (7.07) | 13.5 (12.92)
  Week 52, n=3,6 | 12.7 (20.23) | 22.5 (16.40)

9. Secondary Outcome: VAS Score for Pain
Description: Participants placed a mark on a 0-100 mm VAS to indicate the magnitude of pain, with 0 meaning no pain and 100 meaning the most severe pain.
Time Frame: Baseline (Week 0), Week 2, Week 4, Week 8, Week 12, Week 24, Week 36, Week 52
Population: All enrolled participants who received at least 1 dose of etanercept. Participants analyzed were participants who were evaluated for pain. n=number of evaluable participants at the corresponding visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Number analyzed (Participants) | 65 | 84
mm
  Baseline (Week 0), n=65,84 | 64.8 (19.56) | 60.5 (23.38)
  Week 2, n=42,62 | 42.7 (27.90) | 47.4 (28.63)
  Week 4, n=35,60 | 41.0 (32.31) | 42.7 (31.08)
  Week 8, n=23,47 | 35.2 (38.28) | 41.7 (31.39)
  Week 12, n=16,34 | 35.6 (35.50) | 39.7 (36.57)
  Week 24, n=7,18 | 27.0 (36.52) | 30.0 (30.04)
  Week 36, n=2,13 | 5.0 (7.07) | 20.0 (26.97)
  Week 48, n=3,6 | 13.7 (18.72) | 17.2 (15.09)

10. Secondary Outcome: Number of Participants With Treatment Adherence Rate of 1), <50 Percents (%), 2), >=50% and <70%, 3), >=70% and <80%, 4), >=80% and <100%, 5), >=100% and <120%, and 6), >=120%
Description: Treatment adherence rate was calculated using the following formula: [Actual dosing/expected dosing on the basis of approved product label] × 100%. Counts of participants by 6 levels of treatment adherence rate: 1), <50%, 2), >=50% and <70%, 3), >=70% and <80%, 4), >=80% and <100%, 5), >=100% and <120%, and 6), >=120%.
Time Frame: First day of receiving etanercept up to Week 52
Population: All enrolled participants who received at least 1 dose of etanercept. Participants analyzed were participants who were evaluated for treatment adherence rate; those participants with partial dosing dates were excluded.
Measure: Number; unit: Participants
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Number analyzed (Participants) | 69 | 88
Participants
  <50% | 3 | 3
  >= 50% and <70% | 40 | 44
  >=70% and <80% | 4 | 0
  >=80% and <100% | 4 | 4
  >=100% and <120% | 18 | 36
  >=120% | 0 | 1

11. Secondary Outcome: Evaluate the Association Between Participant's Age and Treatment Adherence Rate
Description: Participants were allocated to 5 groups by age as 10 years separately: <20 years, >=20 and <30 years, >=30 and <40 years, >=40 and <50 years, >50 years. The number of participants with treatment adherence rate 1), <50%, 2), >=50% and <70%, 3), >=70% and <80%, 4), >=80% and <100%, 5), >=100% and <120%, and 6), >=120% were provided for each age group described above.
Time Frame: First day of receiving etanercept up to Week 52
Population: All enrolled participants who received at least 1 dose of etanercept. Participants analyzed were participants who were evaluated for treatment adherence rate; those participants with partial dosing dates were excluded. n=number of evaluable participants at the corresponding age group.
Measure: Number; unit: Participants
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Number analyzed (Participants) | 69 | 88
Participants
  <20 years (<50%), n=3,15 | 1 | 0
  <20 years (>=50% and <70%), n=3,15 | 2 | 11
  <20 years (>=70% and <80%), n=3,15 | 0 | 0
  <20 years (>=80% and <100%), n=3,15 | 0 | 0
  <20 years (>=100% and <120%), n=3,15 | 0 | 4
  <20 years (>=120%), n=3,15 | 0 | 0
  >=20 and <30 years (<50%), n=3,26 | 0 | 1
  >=20 and <30 years (>=50% and <70%), n=3,26 | 3 | 14
  >=20 and <30 years (>=70% and <80%), n=3,26 | 0 | 0
  >=20 and <30 years (>=80% and <100%), n=3,26 | 0 | 2
  >=20 and <30 years (>=100% and <120%), n=3,26 | 0 | 9
  >=20 and <30 years (>=120%), n=3,26 | 0 | 0
  >=30 and <40 years (<50%), n=7,21 | 0 | 0
  >=30 and <40 years (>=50% and <70%), n=7,21 | 3 | 9
  >=30 and <40 years (>=70% and <80%), n=7,21 | 1 | 0
  >=30 and <40 years (>=80% and <100%), n=7,21 | 0 | 1
  >=30 and <40 years (>=100% and <120%), n=7,21 | 3 | 10
  >=30 and <40 years (>=120%), n=7,21 | 0 | 1
  >=40 and <50 years (<50%), n=22,17 | 0 | 1
  >=40 and <50 years (>=50% and <70%), n=22,17 | 13 | 8
  >=40 and <50 years (>=70% and <80%), n=22,17 | 2 | 0
  >=40 and <50 years (>=80% and <100%), n=22,17 | 2 | 1
  >=40 and <50 years (>=100% and <120%), n=22,17 | 5 | 7
  >=40 and <50 years (>=120%), n=22,17 | 0 | 0
  >50 years (<50%), n=34,9 | 2 | 1
  >50 years (>=50% and <70%), n=34,9 | 19 | 2
  >50 years (>=70% and <80%), n=34,9 | 1 | 0
  >50 years (>=80% and <100%), n=34,9 | 2 | 0
  >50 years (>=100% and <120%), n=34,9 | 10 | 6
  >50 years (>=120%), n=34,9 | 0 | 0

12. Secondary Outcome: Number of Participants With Any Abnormal Laboratory Test Results
Description: Number of participants with any abnormal laboratory test results, criteria for abnormalities were complete blood count (CBC) including hemoglobin (<0.8*lower limit of normal[LLN]), mean corpuscular volume (MCV, <0.9*LLN or >1.1*upper limit of normal[ULN]), hematocrit (<0.8*LLN), red blood cell count (<0.8*LLN), platelets (<0.5*LLN or >1.75*ULN), white blood cell count (<0.6*LLN or >1.5*ULN), lymphocytes (<0.8*LLN or >1.2*ULN), neutrophils (<0.8*LLN or >1.2*ULN), basophil (>1.2*ULN), eosinophil (>1.2*ULN), and monocytes (>1.2*ULN); ESR (>1.5*ULN); aspartate aminotransferase (AST,>3.0*ULN); alanine aminotransferase (ALT,>3.0*ULN); blood urea nitrogen (BUN,>1.3*ULN); and creatinine (CRE,>1.3*ULN).
Time Frame: Baseline (Week 0) up to Week 52
Population: All enrolled participants who received at least 1 dose of etanercept. Participants analyzed were participants who were evaluated for laboratory test abnormalities.
Measure: Number; unit: Participants
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Number analyzed (Participants) | 37 | 62
Participants | 25 | 34

13. Secondary Outcome: Tender Joint Count (TJC) for RA Participants
Description: TJC (28 joints) include the joints of shoulders, elbows, wrists, metacarpophalangeal (MCP), proximal interphalangeal (PIP), and the knees. The joints were assessed for tenderness using the following scale: Present (1), Absent (2), Not Done (3), Not Applicable (4). Artificial joints were not assessed.
Time Frame: Baseline (Week 0), Week 2, Week 4, Week 8, Week 12, Week 24, Week 36, Week 52
Population: All enrolled participants who received at least 1 dose of etanercept. Participants analyzed were RA participants who were evaluated for TJC. n=number of evaluable participants at the corresponding visit.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Rheumatoid Arthritis [RA]
Number analyzed (Participants) | 68
Joints
  Baseline (Week 0), n=68 | 10.0 (7.77)
  Week 2, n=44 | 4.0 (4.72)
  Week 4, n=34 | 2.9 (4.02)
  Week 8, n=22 | 1.7 (4.31)
  Week 12, n=17 | 2.0 (4.76)
  Week 24, n=6 | 0.7 (1.21)
  Week 36, n=2 | 0.0 (0.00)
  Week 52, n=3 | 2.0 (1.73)

14. Secondary Outcome: Swollen Joint Count (SJC) for RA Participants
Description: SJC (28 joints) include the joints of shoulders, elbows, wrists, MCP, PIP, and the knees. The joints were assessed for swelling using the following scale: Present (1), Absent (2), Not Done (3), Not Applicable (4). Artificial joints were not assessed.
Time Frame: Baseline (Week 0), Week 2, Week 4, Week 8, Week 12, Week 24, Week 36, Week 52
Population: All enrolled participants who received at least 1 dose of etanercept. Participants analyzed were RA participants who were evaluated for SJC. n=number of evaluable participants at the corresponding visit.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Rheumatoid Arthritis [RA]
Number analyzed (Participants) | 68
Joints
  Baseline (Week 0), n=68 | 5.5 (5.75)
  Week 2, n=44 | 2.3 (3.07)
  Week 4, n=34 | 1.5 (2.54)
  Week 8, n=22 | 0.3 (0.72)
  Week 12, n=17 | 0.5 (0.94)
  Week 24, n=6 | 0.2 (0.41)
  Week 36, n=2 | 0.0 (0.00)
  Week 52, n=3 | 0.3 (0.58)

15. Secondary Outcome: Disease Activity Score (DAS) Based on 28-joints Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR])
Description: DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hour) and PtGA of disease activity on a 0-100 mm VAS: DAS28-4 (ESR)=0.56*square root(TJC 28 joints) + 0.28*square root(SJC 28 joints) + 0.70*ln(ESR) + 0.014*PtGA. DAS28-4 (ESR) above 5.1 indicated high disease activity whereas a DAS28-4 (ESR) below 3.2 indicated low disease activity.
Time Frame: Baseline (Week 0), Week 2, Week 4, Week 12, Week 52
Population: All enrolled participants who received at least 1 dose of etanercept. Participants analyzed were RA participants who were evaluated for DAS28-4 (ESR). n=number of evaluable participants at the corresponding visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis [RA]
Number analyzed (Participants) | 55
units on a scale
  Baseline (Week 0), n=55 | 5.57 (1.338)
  Week 2, n=20 | 4.03 (1.305)
  Week 4, n=18 | 3.31 (1.453)
  Week 8, n=1 | 2.88 (NA) — Standard deviation cannot be calculated since only 1 participant was analyzed at this visit.
  Week 12, n=8 | 2.80 (1.702)
  Week 36, n=1 | 1.20 (NA) — Standard deviation cannot be calculated since only 1 participant was analyzed at this visit.
  Week 52, n=2 | 3.08 (2.083)

16. Secondary Outcome: Number of RA Participants Had DAS28-4 (ESR) Improvement
Description: Counts of participants had good, moderate and no response to treatment with etanercept. Good response was present DAS28-4 (ESR) <=3.2, DAS28-4 (ESR) improvement from baseline >1.2. Moderate response was 1) present DAS28-4 (ESR) >3.2 and <=5.1, DAS28-4 (ESR) improvement from baseline >1.2, or >0.6 and <=1.2; 2) present DAS28-4 (ESR) <=3.2, DAS28-4 (ESR) improvement from baseline >0.6 and <=1.2; or 3) present DAS28-4 (ESR) >5.1, DAS28-4 (ESR) improvement from baseline > 1.2. No response was 1) DAS28-4 (ESR) improvement from baseline <=0.6 regardless present DAS28-4 (ESR), or 2) present DAS28-4 (ESR) >5.1, DAS28-4 (ESR) improvement from baseline >0.6 and <=1.2.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 36, Week 52
Population: All enrolled participants who received at least 1 dose of etanercept. Participants analyzed were participants who were evaluated for DAS28-4 (ESR) improvement. n=number of evaluable participants at the corresponding visit.
Measure: Number; unit: Participants
Arm/Group | Rheumatoid Arthritis [RA]
Number analyzed (Participants) | 17
Participants
  Good response (Week 2), n=17 | 4
  Moderate response (Week 2), n=17 | 10
  No response (Week 2), n=17 | 3
  Good response (Week 4), n=16 | 8
  Moderate response (Week 4), n=16 | 6
  No response (Week 4), n=16 | 2
  Good response (Week 8), n=1 | 1
  Moderate response (Week 8), n=1 | 0
  No response (Week 8), n=1 | 0
  Good response (Week 12), n=7 | 5
  Moderate response (Week 12), n=7 | 2
  No response (Week 12), n=7 | 0
  Good response (Week 36), n=1 | 1
  Moderate response (Week 36), n=1 | 0
  No response (Week 36), n=1 | 0
  Good response (Week 52), n=1 | 1
  Moderate response (Week 52), n=1 | 0
  No response (Week 52), n=1 | 0

17. Secondary Outcome: Number of RA Participants Had Remission of Disease
Description: Counts of participants had remission of disease. Remission of disease was defined by a DAS28-4 (ESR) <2.6.
Time Frame: Baseline (Week 0), Week 2, Week 4, Week 8, Week 12, Week 36, Week 52
Population: All enrolled participants who received at least 1 dose of etanercept. Participants analyzed were participants who were evaluated for DAS28-4 (ESR). n=number of evaluable participants at the corresponding visit.
Measure: Number; unit: Participants
Arm/Group | Rheumatoid Arthritis [RA]
Number analyzed (Participants) | 55
Participants
  Baseline (Week 0), n=55 | 0
  Week 2, n=20 | 2
  Week 4, n=18 | 5
  Week 8, n=1 | 0
  Week 12, n=8 | 4
  Week 36, n=1 | 1
  Week 52, n=2 | 1

ADVERSE EVENTS:
Time Frame: First day of receiving etanercept through the study period until at least 28 after the last dose of etanercept, for SAE, the start time was when the subject provided informed consent or signed data privacy statement.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Rheumatoid Arthritis [RA] | Ankylosing Spondylitis [AS]
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/90
Other Adverse Events (participants affected / at risk) | 8/69 | 9/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis [RA] (N=69) | Ankylosing Spondylitis [AS] (N=90)
Uveitis (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Injection site swelling (General disorders) | 0 | 1
Irritability (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase (Investigations) | 0 | 1
Alanine aminotransferase abnormal (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.